CLINICAL TRIAL: NCT01279564
Title: Comparison Between Etview Tracheoscopic Ventilation Tube - TVT to Standard Endotracheal Intubation During Regular and Difficult Intubation
Brief Title: Comparison Between Etview Tracheoscopic Ventilation Tube - TVT to Standard Endotracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 181-09CTIL; 0181-RMB
Record Dates: First submitted 2011-01-17; First posted 2011-01-19 (Estimated); Results first posted 2014-11-11 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-06

CONDITIONS: Endotracheal Intubation
Keywords: Endotracheal intubation and its outcomes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ETview (Experimental): ETview TVT endotracheal tube
  Interventions: Device: ETview TVT endotracheal tube
- Control (Sham Comparator): Endotracheal tube
  Interventions: Device: Endotracheal tube

INTERVENTIONS:
Device: ETview TVT endotracheal tube — intubation
  Arms: ETview
Device: Endotracheal tube — Intubation
  Arms: Control

SUMMARY:
Airway management is one of the most important tasks facing the physician, especially the anesthesiologist. Fast and correct performance of endotracheal intubations done as normal routine in the operating room, but can save life everywhere.

To make intubation easier, several newly designed tubes and laryngoscopes are developed and tested every year. Their performance is evaluated subjectively by the acting anesthesiologist, and by using objective parameters such as speed of intubation, the force applied during laryngoscopy , or catecholamines secretion during intubation as a stress parameter . The studies set for testing these parameters lead to establish accepted indications for the treatment of the airway in cases of anticipated and unanticipated difficult airway.

In the present study we will compare the performance parameters of intubation using Etview Tracheoscopic Ventilation Tube - TVT to the standard tube, of which most of daily intubations are carried with. The Etview TVT is similar to the standard endotracheal tube; its outer dimensions and material is exactly as the standard tube, the difference is only the inner fiber of the camera.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for elective surgery under general anesthesia with endotracheal intubation

Exclusion Criteria:

* Age under 18 years
* ASA greater than 3
* Lip, oral or airway infection
* Coagulopathy
* Indication to perform Sellick's maneuver for increased risk of aspiration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michal Barak, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult consenting patients that were admitted to Rambam Health Care Campus for laparoscopic sleeve gastrectomy were recruited between February and December 2011
Pre-assignment Details: All recruited patients were enrolled in the study, no one was excluded.
Groups:
- ETview: Endotracheal intubation with ETview TVT
  ETview TVT endotracheal tube: intubation
- Control: Intubation
  Endotracheal tube- standard
Period: Overall Study
Arm/Group | ETview | Control
Started | 40 | 32
Completed | 40 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: Intubation
  Endotracheal tube: Intubation
- Total: Total of all reporting groups
Arm/Group | ETview | Control | Total
Number analyzed (Participants) | 40 | 32 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (4.9) | 42.5 (3.2) | 42.8 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 23 | 49
  Male | 14 | 9 | 23

OUTCOME MEASURES:

1. Primary Outcome: In the Present Study we Will Compare the Performance Parameters of Intubation Using Etview Tracheoscopic Ventilation Tube - TVT to the Standard Tube
Time Frame: 1 year
Reporting Status: Not Posted

2. Primary Outcome: Duration of Endotracheal Intubation
Description: Time between introducing the laryngoscope and inflation of tube's cuff
Time Frame: The induction of general anesthesia, on the operating day (first day)
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- ETview: Endotracheal intubation with ETview TVT
  Duration of intubation
- Control: Intubation
  Duration of intubation
Arm/Group | ETview | Control
Number analyzed (Participants) | 40 | 32
seconds | 29 (10) | 24 (8)

ADVERSE EVENTS:
Time Frame: 1 year
Description: No adverse events
Groups:
- ETview: Endotracheal intubation with ETview TVT
  ETview TVT endotracheal tube: intubation
  No adverse events
- Control: Intubation
  Endotracheal tube: Intubation
  No adverse events
Arm/Group | ETview | Control
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/32
Other Adverse Events (participants affected / at risk) | 0/40 | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ETview (N=40) | Control (N=32)
Difficult intubation or ventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 — Difficulties in introducing the endotracheal tube or ventilating the patient

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less